CLINICAL TRIAL: NCT01096875
Title: Assessment of the Effects of Atorvastatin on Endothelial Progenitor Cells After Coronary ByPass Surgery; A Randomized Controlled Trial
Brief Title: Effects of Atorvastatin on Endothelial Progenitor Cells After Coronary Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara University (Other)
Collaborators: Turkish Society of Hematology (Other)
Responsible Party: Principal Investigator, A. Ruchan Akar, Professor, Consultant Cardiovascular Surgeon, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UMT0043
Record Dates: First submitted 2010-03-16; First posted 2010-03-31 (Estimated); Results first posted 2014-07-09 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Coronary Artery Bypass Surgery; Elective Surgical Procedure
Keywords: Endothelial progenitor cells; Atorvastatin; Coronary surgery
MeSH Terms: interventions — Atorvastatin; ORANGE protein, Arabidopsis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Active Comparator): Hydroxymethylglutaryl-CoA Reductase Inhibitors
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): Atorvastatin like pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — 40mg/day once daily for two weeks prior to surgery
  Other Names: Ator
  Arms: Atorvastatin
Drug: Placebo — 1tb/day once daily for two weeks prior to surgery
  Other Names: Placebo tablets matched to atorvastatin
  Arms: Placebo

SUMMARY:
Experimental data have demonstrated favourable effects of statins on endothelial progenitor cell (EPC) mobilization from the bone marrow, and cardiac homing. The purpose of the present prospective randomized controlled trial is to determine the effects of aggressive atorvastatin treatment (40 mg daily 2-weeks prior to surgery) on the number of endothelial progenitor cells (EPCs) after cardiopulmonary bypass by comparing with placebo.

DETAILED DESCRIPTION:
Endothelial progenitor cells, a subgroup of hematopoietic stem cells have a significant role in vascular homeostasis. In animal models of ischemia, endothelial progenitor cells are rapidly incorporated into sites of neovascularization, have the potential to induce and augment vasculogenesis/ angiogenesis, prevent cardiomyocyte apoptosis in peri-infarct regions, and reduce adverse remodeling. Treatment with atorvastatin has been shown to increase endothelial progenitor cell count in patients with coronary artery disease. Therefore, we will investigate whether atorvastatin augments the number of endothelial progenitor cells after cardiopulmonary bypass in patients undergoing coronary artery bypass surgery (CABG). Thus, we conducted a randomized double-blind, placebo-controlled, 2-way parallel trial in 60 patients undergoing coronary artery bypass surgery. Patients will receive either 2-week treatment with atorvastatin or placebo prior to surgery. Endothelial progenitor cells will be quantitated by flow cytometric phenotyping obtained from peripheral blood samples. In addition, cardiac markers (CK-MB mass, cardiac troponin-I), biochemical profile, liver function tests, high sensitive C-reactive protein (hsCRP) and coagulation profile will be determined at 4 time points: 1) preoperatively (baseline); 2) 6 hours after the end of cardiopulmonary bypass; 3) 24 hours after surgery; 4) 5th days postoperatively. Clinical, operative characteristics, cardiac markers, high sensitive C-reactive protein and endothelial progenitor cell count will be compared between the groups. Adverse outcomes will also be noted and reported.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective isolated coronary artery bypass surgery with on-pump technique
* Written informed consent

Exclusion Criteria:

* Concomitant valve or aortic surgery
* Left ventricular aneurysm repair
* Re-operation
* Emergency surgery
* History of myocardial infarction within less than 4 weeks
* Hepatic impairment
* Chronic renal impairment
* Drug related side effects (allergy or hypersensitivity)
* Familial Hyperlipidemia
* Autoimmune conditions which require steroids

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: RUCHAN AKAR, Assoc. Prof., Study Director — Ankara University Medical Faculty, Department of Cardiovascular Surgery Ankara, Turkey, 06340; ONDER ASLAN, Prof., Study Chair — Ankara University Medical Faculty, Department of Hematology Ankara, Turkey
Locations (1):
- Ankara University Medical Faculty, Department of Cardiovascular Surgery, Ankara, Cebeci, Turkey (Türkiye)

REFERENCES:
- [Derived] Baran C, Durdu S, Dalva K, Zaim C, Dogan A, Ocakoglu G, Gurman G, Arslan O, Akar AR. Effects of preoperative short term use of atorvastatin on endothelial progenitor cells after coronary surgery: a randomized, controlled trial. Stem Cell Rev Rep. 2012 Sep;8(3):963-71. doi: 10.1007/s12015-011-9321-z. PMID 22076751

RESULTS

PARTICIPANT FLOW:
Groups:
- Atorvastatin: Hydroxymethylglutaryl-CoA Reductase Inhibitors
  Atorvastatin : 40mg/day once daily for two weeks prior to surgery
- Placebo: Atorvastatin like pill
  Placebo : 1tb/day once daily for two weeks prior to surgery
Period: Overall Study
Arm/Group | Atorvastatin | Placebo
Started | 30 | 30
Completed | 30 | 29
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 21 | 43
  >=65 years | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (8.6) | 62.2 (8.1) | 61.6 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 19 | 18 | 37
Region of Enrollment [Number; unit: participants]
  Turkey | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Endothelial Progenitor Cells (EPCs) Count (Cells/µl)
Time Frame: Postoperative 6th hours
Measure: Mean (Standard Error); unit: cells/µl
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 30 | 29
cells/µl | 5.00 (0.06) | 2.19 (0.06)

2. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF %) Measured at 30 Days Postoperatively
Time Frame: Change between statin and placebo groups at 30 days postoperatively
Measure: Mean (Standard Deviation); unit: percentage of LVEF
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 30 | 29
percentage of LVEF | 54.3 (7.5) | 53.2 (8.7)

3. Secondary Outcome: High Sensitive C-reactive Protein (hsCRP mg/L)
Time Frame: Postoperative 6th hours
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 30 | 29
mg/L | 72.9 (0.6) | 96.0 (0.7)

4. Secondary Outcome: High Sensitive C-reactive Protein (hsCRP mg/L)
Time Frame: 5 days postoperatively
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 30 | 29
mg/L | 4.3 (0.2) | 11.4 (0.8)

ADVERSE EVENTS:
Time Frame: 30 days postoperatively
Arm/Group | Atorvastatin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/30 | 2/29
Other Adverse Events (participants affected / at risk) | 0/30 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin (N=30) | Placebo (N=29)
Low cardiac output (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The major limitation of this study is lack of functional assessment of EPCs using in vitro analysis of colony forming units because of the financial constraints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes